CLINICAL TRIAL: NCT06400472
Title: A First-in-Human, Phase 1a/1b Trial to Assess the Safety, Tolerability and Preliminary Efficacy of LY4170156, an Antibody-Drug Conjugate Targeting Folate Receptor α-Expressing Tumor Cells, in Participants With Selected Advanced Solid Tumors
Brief Title: A Study of LY4170156 in Participants With Selected Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18863; 2024-511238-11-00 (EU CTIS Number); J5E-OX-JZXA (Other: Eli Lilly and Company); LOXO-FRA-24001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Pancreatic Neoplasm; Colorectal Neoplasms
Keywords: Folate receptor alpha; NSCLC; Ovarian cancer; Cervical cancer; Endometrial cancer; Solid tumor; Lung cancer; Breast cancer; Pancreatic cancer; Colorectal cancer; Anti-drug conjugate; Phase I; Chemotherapy; sofe-m
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms | interventions — Bevacizumab; Carboplatin; Itraconazole; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- LY4170156 (Dose-escalation, Cohort A1) (Experimental): Escalating doses of LY4170156 administered intravenously (IV)
  Interventions: Drug: LY4170156
- LY4170156 (Cohort A1 Parts A and C) (Experimental): LY4170156 administered IV
  Interventions: Drug: LY4170156
- LY4170156 Alone or with Itraconazole. Drug-Drug Interaction (DDI) (Cohort A1: Arm B) (Experimental): LY4170156 administered IV and itraconazole administered orally
  Interventions: Drug: LY4170156; Drug: Itraconazole
- LY4170156 (Dose-optimization, Cohort A2) (Experimental): Comparing 2 or more doses (evaluated during dose escalation) of LY4170156 administered IV
  Interventions: Drug: LY4170156
- LY4170156 (Enrichment Cohort A3) (Experimental): Monotherapy administered IV
  Interventions: Drug: LY4170156
- LY4170156 (Combination Cohort A4) (Experimental): Combination with bevacizumab administered IV
  Interventions: Drug: LY4170156; Drug: bevacizumab
- LY4170156 (Combination Cohort A5) (Experimental): Combination with carboplatin administered IV
  Interventions: Drug: LY4170156; Drug: carboplatin
- LY4170156 Combination with Pembrolizumab (Dose-optimization Cohort A6) (Experimental): Comparing 2 or more doses (evaluated during dose escalation) of LY4170156 administered IV with pembrolizumab
  Interventions: Drug: LY4170156; Drug: pembrolizumab
- LY4170156 (Dose-expansion, Cohort B1-B4) (Experimental): LY4170156 administered IV
  Interventions: Drug: LY4170156

INTERVENTIONS:
Drug: LY4170156 — Intravenous
  Other Names: sofetabart mipitecan
Drug: bevacizumab — IV
  Arms: LY4170156 (Combination Cohort A4)
Drug: carboplatin — IV
  Arms: LY4170156 (Combination Cohort A5)
Drug: Itraconazole — oral
  Arms: LY4170156 Alone or with Itraconazole. Drug-Drug Interaction (DDI) (Cohort A1: Arm B)
Drug: pembrolizumab — IV
  Arms: LY4170156 Combination with Pembrolizumab (Dose-optimization Cohort A6)

SUMMARY:
The purpose of this study is to find out whether the study drug, LY4170156, is safe, tolerable and effective in participants with advanced solid tumors. The study is conducted in two parts - phase Ia (dose-escalation, dose-optimization) and phase Ib (dose-expansion). The study will last up to approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following solid tumor cancers:

  * Dose Escalation: Ovarian (epithelial ovarian, primary peritoneal, and fallopian tube) cancer, endometrial cancer, cervical cancer, non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), pancreatic cancer, or colorectal cancer (CRC)
  * Dose Optimization: Ovarian (epithelial ovarian, primary peritoneal, and fallopian tube) and endometrial cancer
  * Dose Expansion: Low grade serous ovarian cancer, cervical cancer, NSCLC, and TNBC

Exclusion Criteria:

* Individual with known or suspected uncontrolled central nervous system (CNS) metastases
* Individual with history of carcinomatous meningitis
* Individual with active uncontrolled systemic bacterial, viral, fungal, or parasitic infection
* Individual with evidence of corneal keratopathy or history of corneal transplant
* Any serious unresolved toxicities from prior therapy
* Significant cardiovascular disease
* Prolongation of QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 milliseconds (ms)
* History of pneumonitis/interstitial lung disease
* Individuals who are pregnant, breastfeeding or plan to breastfeed during study or within 30 days of last dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: To determine the recommended phase 2 dose (RP2D) of LY4170156 | 1 Cycle (21 days)
  Number of participants with dose-limiting toxicities (DLTs)
Phase 1a: To determine the RP2D or optimal dose of LY4170156 with bevacizumab | 1 Cycle (21 days)
  Number of participants with DLTs
Phase 1a: To determine the RP2D or optimal dose of LY4170156 with carboplatin | 1 Cycle (21 days)
  Number of participants with DLTs
Phase 1a: To determine the RP2D or optimal dose of LY4170156 with pembrolizumab | 1 Cycle (21 days)
  Number of participants with DLTs
Phase 1b: To assess the antitumor activity of LY4170156 Monotherapy: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Up to Approximately 48 Months or 4 Years
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) properties of LY4170156: Minimum Plasma Concentration (Cmin) | First 4 Cycles (84 days)
  PK: Cmin of LY4170156
To characterize the PK properties of LY4170156: Cmin with bevacizumab or carboplatin | First 4 Cycles (Approximately 84 days)
  PK: Cmin of LY4170156
To characterize the PK properties of LY4170156: Cmin with pembrolizumab | First 4 Cycles (84 days)
  PK: Cmin of LY4170156
To characterize the PK properties of LY4170156: Area under the concentration versus time curve (AUC) | First 4 Cycles (84 days)
  PK: AUC of LY4170156
To evaluate the preliminary antitumor activity of LY4170156: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To evaluate the preliminary antitumor activity of LY4170156: Overall response rate (ORR) with bevacizumab or carboplatin or pembrolizumab | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To evaluate the preliminary antitumor activity of LY4170156: Duration of response (DOR) | Up to Approximately 48 Months or 4 Years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Duration of response (DOR) with bevacizumab or carboplatin or pembrolizumab | Up to Approximately 48 Months or 4 Years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Time to response (TTR) | Up to Approximately 48 Months or 4 Years
  TTR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Time to response (TTR) with bevacizumab or carboplatin or pembrolizumab | Up to Approximately 48 Months or 4 Years
  TTR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Progression free survival (PFS) | Up to Approximately 48 Months or 4 Years
  PFS per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Progression free survival (PFS) with bevacizumab or carboplatin or pembrolizumab | Up to Approximately 48 Months or 4 Years]
  PFS per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Disease control rate (DCR) | Up to Approximately 48 Months or 4 Years
  DCR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4170156: Disease control rate (DCR) with bevacizumab or carboplatin or pembrolizumab | Up to Approximately 48 Months or 4 Years
  DCR per investigator assessed RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- United States (9):
  - HonorHealth, Scottsdale, Arizona
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - NYU Langone Health - Long Island, Mineola, New York
  - New York University (NYU) Clinical Cancer Center, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - START Mountain Region, West Valley City, Utah
- Australia (2):
  - Cancer Research SA, Adelaide
  - Icon Cancer Centre South Brisbane, QLD
- France (3):
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de l'Ouest - site St-Herblain, Saint-Herblain
  - Oncopole Claudius Regaud, Toulouse
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Clinico Humanitas, Rozzano
- Japan (3):
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- National Cancer Center, Goyang-si Gyeonggi-do, South Korea
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY4170156 in Participants With Selected Advanced Solid Tumors — https://trials.lilly.com/en-US/trial/482318